CLINICAL TRIAL: NCT00944983
Title: Clinical Validation of the Tiba Medical Ambulo 2400 ABPM According to the ISO 80601-2-30 Standard in Adults, Adolescents, and Children
Status: Completed | Type: Observational
Sponsor: Tiba Medical, Inc. (Industry)
Collaborators: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: UT09-00420-XP
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
Keywords: Hypertension; Hypotension; Clinical Validation; Blood Pressure Accuracy; ISO 81600 Standard; British Hypertension Society; European Society of Hypertension; International Protocol
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Biospecimen Retention: None Retained — Only blood pressure measurements are retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical validation of the Tiba Medical Ambulo 2400 ambulatory blood pressure monitoring system according to the accuracy guidelines of the ISO 80601-2-30 Standard in Adults, Adolescents, and Children.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 3 Years Old

Exclusion Criteria:

* Severe Arrhythmia

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults, Adolescents, and Children of different genders, ages, races & sizes (height, weight & particularly arm size) plus blood pressure ranges (normatensive, hypotensive and hypertensive).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Series of blood pressure measurements obtained in 100+ subjects | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Alpert, MD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Medical Group, Memphis, Tennessee, United States

REFERENCES:
- See also: ISO 80601-2-30 Standard — http://www.iso.org/iso/catalogue_detail.htm?csnumber=44105